CLINICAL TRIAL: NCT06176716
Title: Phase I Clinical Study to Evaluate the Pharmacokinetics, Pharmacokinetics, and Safety of Intravenous Administration of Methoxyethyl Etomidate Hydrochloride for Injection in Subjects With Mild, Moderate, and Normal Hepatic Dysfunction.
Brief Title: Phase 1 Hepatic Insufficiency Trial of Methoxyethyl Etomidate Hydrochloride
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ET-26-HCl-CP-003
Record Dates: First submitted 2023-11-27; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Hepatic Insufficiency
Keywords: Clinical Pharmacology; Hepatic insufficiency
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- participants with mild hepatic impairment (Child-Pugh A) (Experimental)
  Interventions: Drug: ET-26
- participants with moderate hepatic impairment (Child-Pugh B) (Experimental)
  Interventions: Drug: ET-26
- Normal hepatic function (Experimental)
  Interventions: Drug: ET-26

INTERVENTIONS:
Drug: ET-26 — The dose is 0.8 mg/kg, single dose, Infusion time was 60s ± 5s.

SUMMARY:
A Phase I clinical study to compare the pharmacokinetics, pharmacokinetics, and safety of intravenous administration of methoxyetomidate hydrochloride for injection in subjects with mild hepatic insufficiency (Child-pugh A), moderate hepatic insufficiency (Child-Pugh B), and normal hepatic function.Main OBJECTIVE: To evaluate the pharmacokinetic characteristics of metoetomidate hydrochloride for injection in subjects with mild liver dysfunction (Child-Pugh A), moderate liver dysfunction (Child-Pugh B) and normal liver function, and to provide evidence for the clinical application of metoetomidate hydrochloride in patients with liver dysfunction.Secondary objective: To evaluate the safety and pharmacokinetics of metoetomidate hydrochloride for injection in subjects with mild hepatic insufficiency (Child-Pugh A), moderate hepatic insufficiency (Child-Pugh B), and normal hepatic dysfunction.Exploratory objective: To investigate and analyze the relationship between the pharmacokinetic index (MOAA/S, BIS) and the pharmacokinetic parameters of metoetomidate hydrochloride in subjects with different liver function states in this study.The CYP2C19 genotype of the subjects in the study was analyzed, and the influence of gene polymorphism on pharmacokinetic parameters of metoetomidate hydrochloride was explored according to the data of CYP2C19 genotype.The relationship between in vivo exposure to methoxyetomidate hydrochloride and liver injury was analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent before the test, and fully understand the test content, process and possible adverse reactions
2. Be able to complete the study according to the requirements of the test plan 3 Subjects (including partners) were willing to voluntarily use effective contraception from screening until 6 months after the last study drug administration 4 Male or female subjects aged 18-70 years (including cut-off) 5 The weight of male subjects is not less than 50 kg, and the weight of female subjects is not less than 45 kg.Body Mass index (BMI) = weight (kg)/height 2 (m2), BMI in the range of 18-32 kg/m2 (including the threshold) 6 Blood pressure should be between 90-159/60-99 mmHg (including the cutoff);The heart rate should be between 55-100 beats/min (including the critical value);SpO2 suction air should be ≥95% 7 For subjects with normal liver function, normal or abnormal clinical laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function) have no clinical significance 8 No potentially difficult airway (modified Markov score of grade I to II) 9 Subjects with normal liver function had no prior serious primary diseases of major organs, including but not limited to gastrointestinal, respiratory, kidney, liver, nervous, blood, endocrine, tumor, immune, mental, or cardiovascular and cerebrovascular diseases 10 Liver insufficiency with Child-Pugh grade A or B is liver insufficiency due to prior primary liver disease, including but not limited to non-alcoholic steatohepatitis, viral hepatitis (hepatitis B, hepatitis C), etc 11 Patients with liver dysfunction: have not taken medication within 4 weeks prior to screening, or require long-term treatment due to liver disease or other comorbidification and have a stable medication regimen (try to avoid CYP3A4 or CYP2C19 suppressors and strong inducers) 12 Patients with hepatic insufficiency: the glomerular filtration rate eGFR > 60mL/min/1.73m2

Exclusion Criteria:

1. Average daily smoking in the 3 months prior to screening was greater than 5 cigarettes
2. Patients with contraindications to deep sedation/general anesthesia or with a history of sedation/anesthesia accidents
3. Subjects with a history of epilepsy
4. Known to be allergic to methetomidate hydrochloride excipients for injection (mannitol, anhydrous disodium hydrogen phosphate);Or allergy (including drug allergy, allergic disease history, etc.)
5. History of alcohol abuse in the 3 months prior to screening (average daily drinking > 2 units of alcohol (1 unit = 285 mL for beer, or 25 mL for spirits, or 100 mL for wine)
6. History of drug abuse in the 3 months prior to the screening period, or use of benzodiazepines for more than 3 months
7. Donate blood or plasma within 30 days prior to screening, or blood loss ≥200 mL, or plasmapheresis
8. Subjects with normal liver function: Use of any prescription drug or Chinese herbal medicine in the 2 weeks prior to screening other than contraceptives, paracetamol, nonsteroidal anti-inflammatory drugs, local over-the-counter topical preparations
9. Participants who participated in any drug clinical trials within 2 months prior to screening (Participants with liver dysfunction who participated in three or more drug clinical trials within 1 year prior to screening should also be excluded)
10. ECG abnormalities were clinically significant and were judged by the investigator to be unsuitable for participation in the study [if tachycardia/bradycardia, degree II-III atrioventricular block, or prolonged QTcF interval requiring drug therapy (male ≥470 ms, female ≥480 ms),Corrected by Fridericia's formula) or otherwise clinically significant abnormalities determined by the clinician]
11. Female subjects were lactating or had a positive blood pregnancy during the screening period or during the trial
12. Subjects with normal liver function who tested positive for any of the indicators of hepatitis B surface antigen, hepatitis C antibody or hepatitis C core antigen, HIV antigen/antibody or syphilis antibody
13. Patients with serious or clinically significant infections (such as respiratory or central nervous system infections), trauma, or major surgical operations within 4 weeks prior to screening
14. People who were expected to have a tendency to surgery or hospitalization during the trial period
15. People who have consumed any food or beverage containing alcohol (or positive breath test for alcohol), grapefruit/grapefruit juice, methylxanthine (e.g., coffee, tea, cola, chocolate), strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion, etc., in the 1 day prior to administration
16. Urine drug screening positive (morphine, methamphetamine, ketamine, cannabis, ecstasy)
17. People who have used propofol, other sedative/narcotic drugs and/or opioid analgesics or combinations containing analgesics within 72 hours prior to administration
18. Those who had any other factors deemed unsuitable by the investigator for participation in the study
19. Patients with hepatic insufficiency: In addition to the primary liver disease itself, or any clinically significant clinical laboratory test abnormality and/or serious history that the investigator believes may affect the test results, including but not limited to gastrointestinal, respiratory, renal, neurological, hematological, endocrine, immune, psychiatric, or cardiovascular and cerebrovascular diseases
20. patients with liver dysfunction: alpha-fetoprotein > 100 ng/mL;Hemoglobin (Hgb) < 80 g/L, platelet ≤50×109/L;Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥5 times the upper limit of normal (ULN)
21. Patients with liver insufficiency: patients with liver failure, or patients with hepatic encephalopathy, hepatocellular carcinoma (except Barcelona stage 0), esophageal variceal hemorrhage and other complications of cirrhosis that researchers consider inappropriate
22. Patients with liver dysfunction: a history of liver transplantation
23. Patients with liver dysfunction: HIV antigen/antibody screening positive;If syphilis antibody is positive, the rapid plasma rereaction hormone test (RPR) test should be added, and if RPR is also positive, it should be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | up to 5 minutes after infusion
  Cmax
Pharmacokinetic parameters | immediately after infusion to infinite time
  AUC0-inf
Pharmacokinetic parameters | immediately after infusion to 24 hours after infusion
  AUC0-t
Pharmacokinetic parameters | up to 6 hours after infusion
  t1/2

SECONDARY OUTCOMES:
Pharmacodynamic indicators | once within 10 minutes before dosing, once 1 minutes (±5seconds) after dosing, and once 2minutes (±30 seconds) after stopping dosing and during full wakefulness
  MOAA/S score
Pharmacodynamic indicators | 10 minutes before administration to full wakefulness, once every 1 minute
  BIS score

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Study Director — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No